CLINICAL TRIAL: NCT04455334
Title: The Effects of Error-augmented Walking on Gait Performance and Brain Activities in Individuals With Stroke
Brief Title: Error-augmented Walking on Gait Performance and Brain Activities in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202004042RIND
Record Dates: First submitted 2020-06-22; First posted 2020-07-02 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Healthy; Stroke
Keywords: error augmentation,gait symmetry,brain activation,split-belt treadmill,walking adaptation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- healthy (Other): year 1 study
  Interventions: Other: NO INTERVENTION
- stroke (Other): year 1 study
  Interventions: Other: NO INTERVENTION
- active control group (Active Comparator): year 2 study
  Interventions: Other: active control group
- Error-augmented treadmill training (Experimental): year 2 study
  Interventions: Other: Error-augmented treadmill training
- Error-augmented concept combined physical therapy group (Experimental): year 3 study
  Interventions: Other: Error-augmented concept combined physical therapy group
- conventional physical therapy group (Active Comparator): year 3 study
  Interventions: Other: conventional physical therapy group

INTERVENTIONS:
Other: Error-augmented treadmill training — walk on split-belt treadmill
  Arms: Error-augmented treadmill training
Other: active control group — walk on tie-belt treadmill
  Arms: active control group
Other: Error-augmented concept combined physical therapy group — Error-augmented concept combined physical therapy
  Arms: Error-augmented concept combined physical therapy group
Other: conventional physical therapy group — conventional physical therapy
  Arms: conventional physical therapy group
Other: NO INTERVENTION — NO INTERVENTION
  Arms: healthy; stroke

SUMMARY:
This three-year study is proposed to document the effect and further implementation of error-augmented walking on gait performance and brain activities in individuals with stroke. Note that brain activations of post-stroke individuals during locomotion is a relatively unexplored realm. In the first year, study aims to observe the gait performance and brain activity of post-stroke and healthy participants when they walk on the split-belt treadmill, which inputs errors and causing adaptation during locomotion. Second year, study focuses on the long-term effect in aspect of brain activation and gait performance after training the post-stroke individuals with error-augmented treadmill walking. Lastly, study aim to investigate the long-term effect of practically applying the concept of error-augmented training strategy into clinical physical therapy.

The first-year study is a cross-sectional study to recruit post-stroke and healthy participants. Gait performance will be measured by GaitUp system and brain activity during each walking trails will be measured concurrently by functional near infrared spectroscopy (fNIRS). Cadence, stride time, stride length and swing cycle are the gait parameters that will be recorded. Also, symmetry ratio and variability of temporal and spatial parameters will also be calculated. Brain area of interest in this study will be bilateral premotor cortex (PMC), supplementary motor area (SMA) and medial part of primary motor cortex (M1). Study will run one-way analysis of variance (ANOVA) with repeated measures and, if needed, Tukey post hoc test will be used to document the within group and between group differences with p<.05.

The second year and third year study are single-blinded (assessor), randomized controlled trials. In the second year, study will recruit and randomize post-stroke participants into one of the two training groups, error-augmented treadmill training group (ETT group) and active control group (AC group). In ETT group, participants will practice split-belt treadmill walking. And participants in AC group will received traditional treadmill walking. The training duration will be 40 minutes per session, 3 sessions per week for a total of 4 weeks for every group. There will be three evaluations, chronologically, on one day before intervention, one day after completion of intervention and one month after completion of intervention. Gait performance, brain activity, dynamic gait index and sensorimotor ability of lower extremity will be documented. Two-way ANOVA and Tukey post-hoc test will be used to determine the training and follow-up effects with p< .05. During the third year, individuals with stroke will be recruited and randomized to one of the two group, error-augmented concept combined physical therapy group (EAPT group) and conventional physical therapy group (CPT group). Participants in the CPT group will receive thirty-minute conventional physical therapy each session. Instead of training on a split-belt treadmill, participants in EAPT group will receive fifteen-minute walking trainings that implement the error-augmented concept and another fifteen-minute conventional physical therapy each session. The training duration will be 40 minutes per session, 3 sessions per week for a total of 4 weeks for every group. The outcome measurements, and statistical analysis are the same as those described in the second year.

ELIGIBILITY:
The inclusion criteria of stroke participants are

1. first unilateral stroke
2. older than 20 years old
3. medically stable
4. lesion site limited in subcortical area
5. having step length asymmetry (asymmetry ratio ≥ 1.08)
6. ability to walk 10 meters independently without an assistive device.

The inclusion criteria of healthy participants are

1. ability to walk 10 meters independently without an assistive device
2. no any other neurological, psychological, or orthopedic disorders known to interfere the walking performance
3. mini-mental status examination scores > 24 points

The exclusion criteria are

1. Participants who are medical unstable
2. cognitive impaired (mini-mental status examination scores < 24 points)
3. diagnosed with other neurological, psychological, or orthopedic disorders known to interfere the participation to the study
4. with the diagnosis which the contraindication includes exercise

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2023-06-03 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of walking performance - Cadence | Change from Baseline cadence at 4 weeks
  The unit is steps per minutes
Change of walking performance - Cadence | Change from Baseline cadence at 8 weeks
  The unit is steps per minutes
Change of walking performance - stride time | Change from Baseline cadence at 4 weeks
  The unit is seconds
Change of walking performance - stride time | Change from Baseline cadence at 8 weeks
  The unit is seconds
Change of walking performance - stride length | Change from Baseline cadence at 4 weeks
  The unit is cm
Change of walking performance - stride length | Change from Baseline cadence at 8 weeks
  The unit is cm
Change of walking performance - swing cycle | Change from Baseline cadence at 4 weeks
  The unit is percentage (%)
Change of walking performance - swing cycle | Change from Baseline cadence at 8 weeks
  The unit is percentage (%)
Change of walking performance - symmetry ratio | Change from Baseline cadence at 4 weeks
  V(larger value) / V(lesser value), V=step length(spatial) or step time(temporal)
Change of walking performance - symmetry ratio | Change from Baseline cadence at 8 weeks
  V(larger value) / V(lesser value), V=step length(spatial) or step time(temporal)
Change of walking performance - variability | Change from Baseline cadence at 4 weeks
  CV(coefficient of variation) = standard deviation/mean x 100% of the stride length(spatial) or stride time(temporal)
Change of walking performance - variability | Change from Baseline cadence at 8 weeks
  CV(coefficient of variation) = standard deviation/mean x 100% of the stride length(spatial) or stride time(temporal)

SECONDARY OUTCOMES:
Brain activities over premotor cortex | Change from Baseline cadence at 4 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over premotor cortex | Change from Baseline cadence at 8 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over supplementary motor area | Change from Baseline cadence at 4 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over supplementary motor area | Change from Baseline cadence at 8 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over primary motor cortex | Change from Baseline cadence at 4 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.
Brain activities over primary motor cortex | Change from Baseline cadence at 8 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) is used to detect the hemodynamics.

OTHER OUTCOMES:
Dynamic Gait Index | Change from Baseline cadence at 4 weeks
Dynamic Gait Index | Change from Baseline cadence at 8 weeks
Fugl-Meyer assessment | Change from Baseline cadence at 4 weeks
  Sensorimotor impairment of lower extremity
Fugl-Meyer assessment | Change from Baseline cadence at 8 weeks
  Sensorimotor impairment of lower extremity

CONTACTS AND LOCATIONS:
Overall Officials: Yanci Liu, Ph.D, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan